CLINICAL TRIAL: NCT04107090
Title: Role of Lung Ultrasound In Assessment Of Recruitment Maneuvers In Ventilated Preterms With Respiratory Distress Syndrome and Its Correlation With Tracheal IL-6 Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Reda Fikry Kamel, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Lung Ultrasound
Record Dates: First submitted 2019-09-19; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Intervention Model Description: The study was conducted on 44 preterm neonates who were mechanically ventilated for respiratory distress syndrome (RDS). Then they were allocated randomly to one of 2 groups in order by admission:
  Group A: it included 22 patients on whom the recruitment manoeuvre was applied guided by lung ultrasonography.
  Group B: it included 22 patients on whom the recruitment maneuver was not ultrasound guided. This is considered the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US guided lung recruitment (Experimental): Group A: it included 22 patients on whom the recruitment manoeuvre was applied guided by lung ultrasonography.
  Interventions: Other: lung recruitment maneuver; Other: tracheal IL-6 level; Other: US guided lung recruitment maneuver
- Non US guided lung recruitment (Other): Group B: it included 22 patients on whom the recruitment maneuver was not ultrasound guided. This is considered the control group.
  Interventions: Other: lung recruitment maneuver; Other: tracheal IL-6 level

INTERVENTIONS:
Other: lung recruitment maneuver — Lung recruitment maneuver done for ventilated preterm neonates diagnosed with respiratory distress syndrome
Other: tracheal IL-6 level — tracheal IL-6 level was measured before and after recruitment maneuver
Other: US guided lung recruitment maneuver — Lung recruitment maneuver done for ventilated preterm neonates diagnosed with respiratory distress syndrome guided by lung ultrasound
  Arms: US guided lung recruitment

SUMMARY:
This work is designed to:

1. Evaluate the efficacy of lung ultrasonography in detecting opening and closing lung pressures in ventilated preterm neonates with respiratory distress syndrome.
2. Determine the efficacy of lung ultrasonography in optimizing lung volume and its correlation with pulmonary inflammatory reaction as evidenced by IL-6 level in tracheal aspirate.

DETAILED DESCRIPTION:
The studied population included 44 preterm infants. Anthropometric measurements, gestational age, sex, mode of delivery, maternal disease and Apgar score were found to be matched in the two studied groups indicating successful randomization as seen in these balanced demographic variables between the groups.

The studied population included 44 preterm infants. Then they were allocated randomly to one of 2 groups in order by admission:

Group A: included 22 patients on whom the recruitment maneuver was applied guided by lung ultrasonography.

Group B: included 22 patients on whom the recruitment maneuver was not ultrasound guided. This is considered the control group.

Anthropometric measurements, gestational age, sex, mode of delivery, maternal disease and Apgar score were found to be matched in the two studied groups indicating successful randomization as seen in these balanced demographic variables between the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age ≤ 36 weeks.
2. In need for invasive mechanical ventilation for RDS according to Downes Score .

Exclusion Criteria:

* excluded:

  1. Major upper or lower airway anomalies.
  2. Significant congenital anomalies including cardiac, abdominal or respiratory.
  3. Surgical cases
  4. Inborn errors of metabolism
  5. Early onset sepsis.
  6. Meconium aspiration syndrome.
  7. Hypoxic ischemic encephalopathy.

Ages: 1 Hour to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Lung ultrasound and diagnosis of respiratory distress syndrome | 1 year
  Forty four preterm neonates diagnosed with respiratoey distress syndrome had lung ultrasound assessment . Its grading was N=normal (presence of lung sliding with A lines or fewer than two isolated B lines) , B1=multiple well-defined B lines , B2=multiple coalescent B lines , C=Consolidation.
Lung ultrasound and recruitment maneuver | 1 year
  An ultrasound re aeration score is calculated from changes in the ultrasound pattern of each region examined during the recruitment maneuver (N,B1,B2,C).
Lung ultrasound guided recruitment maneuver and the period of oxygen dependency. | 1 year
  The relation between early lung recruitment maneuver guided by lung ultrasound and how many days requiring oxygen therapy in the NICU .
Lung ultrasound guided recruitment maneuver and the total number of NICU admission days. | 1 year
  The relation between early lung recruitment maneuver guided by lung ultrasound and how many days requiring admission in the NICU .
Lung ultrasound guided recruitment maneuver and its relation to lung inflammation | 1 year
  Tracheal aspirate IL-6 is measured initially before recruitment maneuver, and on the third day if still ventilated ,or before extubation if done earlier than the third day.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Univeristy, Cairo, Egypt